CLINICAL TRIAL: NCT04751175
Title: Ketamine and Dexametasone in the Management of Pain in Lumbar Arthrodesis
Brief Title: Management of Pain in Lumbar Arthrodesis
Acronym: KETASONA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Principal Investigator, Dr Emili Leon, Principal Investigator, Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EudraCT number 2012-002518-38
Record Dates: First submitted 2020-08-06; First posted 2021-02-12 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketamine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Single-center, controlled, prospective and randomized clinical trial, phase IV, to determine the effect of perioperative intravenous administration of ketamine and dexamethasone in patients undergoing lumbar arthrodesis
Who Masked: Participant, Investigator
Masking Description: To preserve the masking of the study, the randomization system has been carried out by the pharmacy service personnel using the EPIDAT 4.0 program and only the personnel responsible for the pharmacy will know the randomization tables and codes. The main investigator will have the emergency codes in case of need by contacting the pharmacy service
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ketamina bolus plus Dexamethasone bolus plus infusion ketamine (Experimental): Ketamine bolus (0.5 mg / kg) + dexamethasone 0.1 mg / kg bolus + ketamine infusion (0.1 mg / kg / h) up to three hours after admission to the Post-Anesthesia Resuscitation Unit (URPA)
  Interventions: Drug: Ketamine; Drug: Dexamethasone
- Ketamine bolus plus ketamine infusion (Experimental): Ketamine bolus (0.5 mg / kg) + physiological serum bolus + ketamine infusion (0.1 mg / kg / h) up to three hours after admission to the URPA.
  Interventions: Drug: Ketamine; Drug: Physiologic saline
- Dexametasone arm (Active Comparator): Saline bolus + dexamethasone bolus 0.1 mg / kg + saline infusion up to three hours after admission in URPA
  Interventions: Drug: Dexamethasone; Drug: Physiologic saline
- Saline bolus (Placebo Comparator): Saline bolus + saline bolus + saline infusion up to three hours after admission to the URPA
  Interventions: Drug: Physiologic saline

INTERVENTIONS:
Drug: Ketamine — Ketamine, being a non-competitive antagonist of NMDA receptors, could represent a good option as an opioid treatment enhancer for acute postoperative pain and avoid chronic pain, by reducing the '' wind-up '' phenomenon of central sensitization
  Arms: Ketamina bolus plus Dexamethasone bolus plus infusion ketamine; Ketamine bolus plus ketamine infusion
Drug: Dexamethasone — A meta-analysis published in September 2011 affirms that the administration of dexamethasone at a dose of 0.1 mg / kg is an effective complement to multimodal analgesia strategies to reduce postoperative pain and opioid consumption after surgery.
  Preoperative administration of the drug produces a more consistent analgesic effect than intraoperative administration
  Arms: Dexametasone arm; Ketamina bolus plus Dexamethasone bolus plus infusion ketamine
Drug: Physiologic saline — placebo
  Arms: Dexametasone arm; Ketamine bolus plus ketamine infusion; Saline bolus

SUMMARY:
KETAMINE AND DEXAMETASONE IN THE MANAGEMENT OF PAIN IN LUMBAR ARTHRODESISPhase IV prospective randomized controlled single-center clinical trial to determine the effect of intravenous ketamine and dexamethasone administration perioperatively in patients undergoing lumbar arthrodesis.

DETAILED DESCRIPTION:
The need to carry out this study is to evaluate the analgesic effects after the administration of ketamine and dexamethasone intravenously perioperatively in patients undergoing lumbar arthrodesis and, likewise, study the incidence of pain and protocolize perioperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age> 18 years
* ASA I-III.
* Lumbar arthrodesis.
* Patients who have signed the preoperative informed consent for participation in the study.

Exclusion Criteria:

* Unstable coronary heart disease
* Glaucoma
* History of allergy to ketamine, dexamethasone, or morphic chloride
* Dementia or inability to understand IC and study
* Pluricomplicated diabetes mellitus difficult to control
* Patients who have taken an experimental drug 30 days before the start of the study or who are included in any type of study of an experimental drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2013-07-04 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Morphic Chloride (PCA) to treat pain during the post-operative period. Consumption of morphics will be evaluated | 4 hours post operative
  Consumption of morphics

SECONDARY OUTCOMES:
Incidence of postoperative nausea and vomiting (PONV). | 4 hours post operative
  Incidence of postoperative nausea and vomiting
Efficay of study treatment regarding pain at 3 postoperative months | 3 months
  Pain at 3 postoperative months assessed by EVA scale pain. This is a visual analogue scale regarding pain.It consists of a 10-centimeter horizontal line, at the ends of which are the extreme expressions of a symptom. In the left is the absence or less intensity and in the right the greater intensity. The patient is asked to mark on the line the point that indicates the intensity and measure it with a millimeter ruler. The intensity is expressed in centimeters or millimeters. The evaluation will be: 1.Mild pain if the patient scores pain less than 3. 2.Moderate pain if the evaluation is between 4 and 7. 3.Severe pain if the evaluation is equal to or greater than 8.
Adverse side effects:Hallucinations / Delirium.Sedation. Diplopia, Hyperglycemia Respiratory depression (Sat <90%) | 4 hours post operative
  Rate of patients that presented adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Emili Leon, MD, Principal Investigator — Hospital Dr Josep Trueta and Hospital Santa Caterina
Locations (1):
- Hospital Dr Josep Trueta, Girona, Spain